CLINICAL TRIAL: NCT05390112
Title: Cohort Study of Patients With Hepatocellular Carcinoma and Circulating Tumor DNA Monitoring of Chemoembolization
Acronym: Mona-Lisa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/330/OB
Record Dates: First submitted 2022-05-09; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Circulating Tumor DNA; Hepatocellular Carcinoma Non-resectable; Transarterial Chemoembolization
Keywords: cell-free DNA; circulating tumor DNA; hepatocellular carcinoma;
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cfDNA ; ctDNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: DNA — ctDNA; cfDNA

SUMMARY:
Cohort study to assess the impact of ctDNA detection in the follow-up and management of patients with hepatocellular carcinoma treated by TACE

DETAILED DESCRIPTION:
The incidence of hepatocellular carcinoma (HCC) has increased significantly over the past 30 years.

The majority of HCCs present at an intermediate stage, ineligible for a curative surgical approach and the reference treatment in this situation corresponds to a palliative locoregional treatment of Transarterial chemoembolization (TACE). This treatment modality can be repeated several times and the interval between each session as well as the modalities to evaluate the efficacy of this procedure remain poorly codified. This evaluation is currently based on imaging performed at one month (M1) (MRI and/or CT scan) more or less associated with the study of the variation of the alphafetoprotein level measured before (baseline) and after (M1) the treatment. However, these evaluation tools have many limitations and remain imperfect in predicting response to treatment.

In this context, liquid biopsy, which is experiencing significant growth in oncology, could be a promising tool. It is characterized by the detection of tumor elements in the bloodstream such as circulating tumor DNA (ctDNA). Several studies have successfully demonstrated the diagnostic or prognostic value of ctDNA in patients followed for HCC.

the aim of our study is to evaluate the impact of ctDNA detection in the follow-up of patients treated by TACE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HCC diagnosed on consensus radiological criteria in cirrhotic patients (EASL-EORTC 2012): helical CT or MRI with triple arterial, portal, and late acquisition. The diagnosis is based on the presence of hypervascularization at the early arterial time (wash-in) with wash-out (hypodensity or hypointensity compared with non-tumor liver parenchyma) at the portal phase or late phase compared with non-tumor parenchyma.
* Histologically diagnosed HCC in the absence of an imaging diagnosis
* Patient with a first TACE (naive) or not, regardless of the number of previous procedures
* Patient naïve or on a new line of oncological treatment, regardless of the number of previous lines of treatment.
* Treatment decision validated by the digestive oncology staff.
* Patient having read and understood the information letter and signed the informed consent.
* Patient follow-up performed at the Charles Nicolle University Hospital in Rouen.

Exclusion Criteria :

* Other active cancer or hematological malignancy, currently being treated
* Patient not affiliated to the social security system
* Pregnant woman or woman in labour or breastfeeding
* Person deprived of liberty by an administrative or judicial decision
* Person placed under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patient with a first TACE (naive) or not, regardless of the number of previous procedures
  * Patient naïve or on a new line of oncological treatment, regardless of the number of previous lines of treatment.
Sampling Method: Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiological response at 1 month according to mRECIST and ctDNA detection | 4 to 6 weeks
  radiological response : mRECIST (progressive disease; stable disease, partial response, complete response) LIRADS (LR-TR Nonviable, LR-TR Equivocal, LR-TR Viable); ctDNA at 1 month detection (yes or no)

SECONDARY OUTCOMES:
Progression-free survival and overall survival | 4 to 6 weeks
  progression-free Survival and overall Survival (months)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent VERDIER, MD, Principal Investigator — vincent.verdier@chu-rouen.fr
Locations (1):
- CHU de Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No